CLINICAL TRIAL: NCT04055012
Title: Metformin and Beyond: Individualizing Care for Low Back Pain
Brief Title: Effects of Metformin on Low Back Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding closed.
Sponsor: Gwendolyn Sowa (Other)
Responsible Party: Sponsor-Investigator, Gwendolyn Sowa, Professor and Chair Department of Physical Medicine and Rehabilitation, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY19010007
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Metformin; Placebo
MeSH Terms: conditions — Low Back Pain | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- High Dose Metformin (Experimental): High Dose Metformin Group (n=100). Subjects will receive metformin and will be instructed to take 2 tabs per day (1,000mg) for the first week then increase to 3 tabs per day (1,500mg) for the remaining 6 months.
  Interventions: Drug: Metformin
- Low Dose Metformin (Experimental): Low Dose Metformin Group (n=100). Subjects will receive metformin and will be instructed to take 1 tab per day (1 metformin tab (500mg) for 6 months.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo Group (n=100). Subjects will receive placebo and will be instructed to take either 2 tabs per day for the first week then increase to 3 tabs per day for the remaining 6 months OR take 1 placebo tab for 6 months.
  Interventions: Drug: Placebo
- Wait-List Control (Other): Control Group (n=100). Subjects will be told that they are in the wait-list control group. They will have a 3 month "waiting period" before they will be randomized again to a treatment group. They will be randomized to one of the previous groups.
  Interventions: Drug: Metformin; Drug: Placebo

INTERVENTIONS:
Drug: Metformin — 500mg tabs of Metformin Extended Release
  Other Names: Glucophage; Glucophage Extended Release; Metformin Extended Release; Metformin ER
  Arms: High Dose Metformin; Low Dose Metformin; Wait-List Control
Drug: Placebo — Placebo Tabs
  Arms: Placebo; Wait-List Control

SUMMARY:
The purpose of the current study is to determine the effects of metformin in non-diabetic patients with low back pain, and identify novel targets for future treatments

DETAILED DESCRIPTION:
Outcome measures were updated after the initial submission to clinicaltrials.gov. The outcomes were changed in the Institutional Review Board protocol but not updated on clinicaltrials.gov. These outcome measures have since been updated to reflect what was collected for the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Diagnosed with axial low back pain (low back pain more severe than pain in other parts of the body, without radiation of pain into the lower extremities).
* Women of child bearing potential must have a negative serum pregnancy test at baseline.

Exclusion Criteria:

* Diagnosed with rheumatoid arthritis, lupus, other autoimmune/systemic inflammatory arthropathies
* Progressive lower extremity weakness or numbness
* Recent oral steroid use (within last 3 months)
* NSAID use
* Chronic kidney disease (eGFR <60)
* Diagnosis of diabetes mellitus
* Subjects must not be pregnant or breastfeeding, or planning to become pregnant or breastfeed during the course of the trial
* Unable to take an oral medication in a non crushable pill form
* Taking metformin presently or within the last 6 months
* History of allergy to metformin
* History of lactic acidosis
* Severe Hepatic dysfunction
* Currently taking a diabetic medication such as sitagliptin, saxagliptin, linagliptin, alogliptin, sitagliptin with metformin
* Currently taking a Carbonic anhydrase inhibitor such as topiramate, zonisamide, acetazolamide, dichlorphenamide, methazolamide
* Currently taking cimetidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Sowa, MD, PhD, Principal Investigator — The University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Kaufmann Medical Building, Pittsburgh, Pennsylvania
  - UPMC Wexford Spine Center, Wexford, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose Placebo: High Dose Placebo Group (n=50). Subjects will receive placebo and will be instructed to take 2 tabs per day for the first week then increase to 3 tabs per day for the remaining 6 months.
  Placebo: Placebo Tabs
- Low Dose Placebo: Low Dose Placebo Group (n=50). Subjects will receive placebo and will be instructed to take 1 placebo tab for 6 months.
  Placebo: Placebo Tabs
Period: Overall Study
Arm/Group | High Dose Metformin | Low Dose Metformin | High Dose Placebo | Low Dose Placebo
Started | 8 (2 participants were from wait-list control group) | 8 (1 participant was from wait-list control group) | 4 (1 participant was from wait-list control group) | 3
Completed | 6 | 4 | 2 | 3
Not Completed | 2 | 4 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 1 | 0
Not completed — Metformin Recall | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Metformin | Low Dose Metformin | High Dose Placebo | Low Dose Placebo | Total
Number analyzed (Participants) | 8 | 8 | 4 | 3 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 4 | 3 | 21
  >=65 years | 2 | 0 | 0 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (16.31826321) | 48 (11.86155254) | 42 (20.82266393) | 45 (16.19670748) | 47 (14.83639367)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 2 | 3 | 18
  Male | 2 | 1 | 2 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 8 | 4 | 2 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 0 | 1 | 5
  White | 5 | 7 | 3 | 2 | 17
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 4 | 3 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Numeric Pain Rating Scale
Description: Scores range from 0 to 10 with a higher score indicating more severe pain
Time Frame: Up to 15 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Dose Metformin | Low Dose Metformin | High Dose Placebo | Low Dose Placebo
Number analyzed (Participants) | 6 | 4 | 2 | 3
score on a scale
  change in pain score | -1.16 (0.98) | -1.5 (0.58) | -1.5 (0.71) | 0.33 (3.06)
  baseline pain score | 5.33 (1.03) | 5.75 (2.22) | 6 (2.83) | 2.33 (2.08)

2. Primary Outcome: Change From Baseline in Oswestry Disability Index (ODI)
Description: Scores range from 0% to 100% with higher scores indicating greater disability
Time Frame: Up to 15 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Low Dose Placebo: Low Dose Placebo Group (n=100). Subjects will receive placebo and will be instructed to take 1 placebo tab for 6 months.
  Placebo: Placebo Tabs
Arm/Group | High Dose Metformin | Low Dose Metformin | High Dose Placebo | Low Dose Placebo
Number analyzed (Participants) | 6 | 4 | 2 | 3
score on a scale
  average ODI change | -3 (7.01) | -2.5 (12.37) | -8 (2.83) | -8.67 (10.07)
  baseline ODI | 23.33 (4.13) | 26 (9.38) | 21 (1.41) | 20.67 (10.26)

3. Secondary Outcome: Change From Baseline in BACPAC (Back Pain Consortium) Minimum Dataset: Pain Outcomes Assessment
Description: Current pain on average reported on 0-10 scale, higher scores indicate greater pain
Time Frame: Up to 15 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Dose Metformin | Low Dose Metformin | High Dose Placebo | Low Dose Placebo
Number analyzed (Participants) | 6 | 4 | 2 | 3
score on a scale | -1.33 (1.21) | -1.5 (1) | 0.5 (0.71) | -0.33 (1.15)

4. Secondary Outcome: Change From Baseline in 10 Meter Walk Test
Description: Subject is timed walking at self-selected speed. A faster time (fewer seconds to complete the walk) is associated with better outcome.
Time Frame: Up to 15 months
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- High Dose Placebo: Placebo Group (n=50). Subjects will receive placebo and will be instructed to take 2 tabs per day for the first week then increase to 3 tabs per day for the remaining 6 months.
  Placebo: Placebo Tabs
Arm/Group | High Dose Metformin | Low Dose Metformin | High Dose Placebo | Low Dose Placebo
Number analyzed (Participants) | 6 | 4 | 2 | 3
seconds | -2.71 (5.26) | -0.57 (1.91) | -0.73 (0.47) | -0.05 (1.26)

5. Secondary Outcome: Change From Baseline in Fear Avoidance Questionnaire
Description: Scores range from 0 to 96 in which a higher score indicates greater fear avoidance beliefs
Time Frame: Up to 15 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Dose Metformin | Low Dose Metformin | High Dose Placebo | Low Dose Placebo
Number analyzed (Participants) | 6 | 4 | 2 | 3
score on a scale | -1.67 (5.20) | -0.25 (8.81) | -7 (4.24) | -5.67 (3.79)

6. Secondary Outcome: Change From Baseline in STarT Back Tool
Description: Scores range from 0-9. A higher score indicates higher risk of persisting disabling symptoms.
Time Frame: Up to 15 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Dose Metformin | Low Dose Metformin | High Dose Placebo | Low Dose Placebo
Number analyzed (Participants) | 6 | 4 | 2 | 3
score on a scale | -1.83 (2.40) | -0.5 (1.29) | 0 (2.83) | -0.33 (3.06)

7. Secondary Outcome: Change From Baseline in 6-item Pain Catastrophizing Scale
Description: Score range from 0 to 24 with a higher score indicating a higher degree of catastrophizing
Time Frame: Up to 15 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Dose Metformin | Low Dose Metformin | High Dose Placebo | Low Dose Placebo
Number analyzed (Participants) | 6 | 4 | 2 | 3
score on a scale | -1.67 (3.88) | 0.75 (4.79) | -2 (1.41) | 0.33 (3.79)

8. Secondary Outcome: Change From Baseline in Positive Outlook v1.0 - Short Form 6a
Description: For most PROMIS domains, a score of 50 is the average for the United States general population with a standard deviation of 10 because calibration testing was performed on a large sample of the general population. A higher score indicates a more positive outlook.
Time Frame: Up to 15 months
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | High Dose Metformin | Low Dose Metformin | High Dose Placebo | Low Dose Placebo
Number analyzed (Participants) | 6 | 4 | 2 | 3
T score | -1.9 (5.78) | 0.225 (5.97) | -2.55 (1.20) | -10.27 (20.35)

9. Secondary Outcome: Change From Baseline in PROMIS (Patient-Reported Outcomes Measurement Information System) 29
Description: The PROMIS (Patient-Reported Outcomes Measurement Information System) 29 is a 29 question assessment of 8 domains of health related quality of life (physical function, fatigue, sleep disturbance, pain interference, anxiety, depression, ability to participate in social roles and activities, and cognitive function. For most PROMIS domains, a score of 50 is the average for the United States general population with a standard deviation of 10 because calibration testing was performed on a large sample of the general population. Higher T scores indicates greater report of the concept being measured.
Time Frame: Up to 15 months
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | High Dose Metformin | Low Dose Metformin | High Dose Placebo | Low Dose Placebo
Number analyzed (Participants) | 6 | 4 | 2 | 3
T score
  Change from baseline in Physical function | -0.62 (4.26) | -2.075 (3.089) | -0.6 (9.48) | -1.43 (2.48)
  Change from baseline in Anxiety | 0.55 (5.32) | -3.075 (3.27) | -6.75 (1.34) | -6.63 (5.75)
  Change from baseline in Depression | 2.25 (6.97) | 2.3 (5.72) | -1.35 (5.87) | -7.8 (8.17)
  Change from baseline in Fatigue | -1.35 (12.90) | -3.2 (6.4) | -0.85 (6.72) | 0.43 (6.36)
  Change from baseline in Sleep disturbance | 1 (4.76) | 0.275 (3.24) | -1.2 (5.66) | -1.33 (1.40)
  Change from baseline in Ability to participate in social roles and activities in the past 7 days | -3.1 (6.44) | -1.575 (9.45) | -3.5 (4.95) | 1.27 (2.19)
  Change from baseline in Pain interference in the past 7 days | -1.55 (3.22) | -4.175 (7.40) | -4.8 (1.70) | 3.07 (5.31)
  Change from baseline in Cognitive function-Abilities | 0 (13.28) | 0 (6.70) | -6.75 (3.61) | -1.07 (1.85)

10. Secondary Outcome: Change From Baseline in General Self-Efficacy - Short Form 4a
Description: For most PROMIS domains, a score of 50 is the average for the United States general population with a standard deviation of 10 because calibration testing was performed on a large sample of the general population. A higher score indicate higher self efficacy.
Time Frame: Up to 15 months
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | High Dose Metformin | Low Dose Metformin | High Dose Placebo | Low Dose Placebo
Number analyzed (Participants) | 6 | 4 | 2 | 3
T score | -3.97 (8.01) | -0.65 (3.90) | 5.45 (7.71) | -8.2 (9.63)

11. Secondary Outcome: Change From Baseline in Global Physical Activity Questionnaire
Description: This questionnaire developed by the World Health Organization measures physical activity at work or school, household, travel, recreational and sedentary behaviors, measured in MET (metabolic equivalent)-minutes per week (continuous variable).
Time Frame: Up to 15 months
Measure: Mean (Standard Deviation); unit: MET- minutes per week
Arm/Group | High Dose Metformin | Low Dose Metformin | High Dose Placebo | Low Dose Placebo
Number analyzed (Participants) | 6 | 4 | 2 | 3
MET- minutes per week | -1100 (3325.9) | -1825 (2953.0) | 1050 (551.54) | -277.33 (240.71)

12. Secondary Outcome: Change From Baseline in McGill Pain Questionnaire
Description: Scores range from 0 to 45 with a higher score indicating more qualitatively severe and impactful pain.
Time Frame: Up to 15 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Dose Metformin | Low Dose Metformin | High Dose Placebo | Low Dose Placebo
Number analyzed (Participants) | 6 | 4 | 2 | 3
score on a scale | -4.83 (3.43) | -2.5 (5.80) | -3.5 (2.12) | -11.67 (19.86)

13. Secondary Outcome: Change in Charlson Comorbidity Index
Description: Measures overall health with a higher score more likely predicative of mortality or higher resource use. Scale is scored 0-37.
Time Frame: Up to 15 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Dose Metformin | Low Dose Metformin | High Dose Placebo | Low Dose Placebo
Number analyzed (Participants) | 6 | 4 | 2 | 3
score on a scale | 0.17 (0.41) | 0.25 (0.5) | 0 (0) | 0 (0)

14. Secondary Outcome: Change From Baseline in Financial Strain
Description: Measures strain of finances. Score ranges from 1-4. The lower the score the harder the financial strain.
Time Frame: Up to 15 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Dose Metformin | Low Dose Metformin | High Dose Placebo | Low Dose Placebo
Number analyzed (Participants) | 6 | 4 | 2 | 3
score on a scale | -0.16 (0.98) | 0 (0) | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: up to 15 months
Arm/Group | High Dose Metformin | Low Dose Metformin | High Dose Placebo | Low Dose Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 6/8 | 6/8 | 2/2 | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Metformin (N=8) | Low Dose Metformin (N=8) | High Dose Placebo (N=2) | Low Dose Placebo (N=3)
Abnormal Lab Value - Low Vitamin B12 (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abnormal Lab Value - Elevated ESR (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abnormal Lab Value - Low Alkaline Phosphatase (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal Lab Value - Hypoglycemia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abnormal Lab Value - Elevated CBC (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal Lab Value - Hypercalcemia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal Lab Value - Elevated Potassium (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low Iron (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Acid Reflux (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gas (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Cramping (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 4 (5) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was halted early due to funding redirection. Due to limited sample size, formal statistical analysis for between group comparisons was not feasible, and no clear trends were established.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT04055012/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-11): https://cdn.clinicaltrials.gov/large-docs/12/NCT04055012/SAP_001.pdf
  • Informed Consent Form (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT04055012/ICF_002.pdf